CLINICAL TRIAL: NCT03093246
Title: Evaluation of Omega-3 Polyunsaturated Fatty Acids Plus Low-dose Aspirin Daily Supplementation in Non-surgical Therapy to Treat Generalized Aggressive Periodontitis: Randomized Controlled Clinical Trial
Brief Title: Omega-3 Plus Low-dose Aspirin Daily Supplementation in Non-surgical Therapy to Treat Aggressive Periodontitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, PhD Adjunt professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HMT+UPD CFA
Record Dates: First submitted 2017-03-22; First posted 2017-03-28 (Actual); Results first posted 2021-07-29 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-12

CONDITIONS: Aggressive Periodontitis
Keywords: Full-mouth ultrasonic debridement; Aspirin; Omega-3 polyunsaturated fatty acids; Non-surgical therapy
MeSH Terms: conditions — Aggressive Periodontitis | interventions — Docosahexaenoic Acids; Fish Oils; Aspirin; Periodontal Debridement

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Placebo Comparator): In this group (n = 19), patients will take placebo pills and full-mouth ultrasonic debridement will be performed to treat diseased sites.
  Interventions: Other: Placebo; Procedure: Full-mouth ultrasonic debridement
- Test Group (Experimental): In this group (n = 19), patients will take 3 g of omega-3 polyunsaturated fatty acids and 100 mg of aspirin daily over a period of 180 days and full-mouth ultrasonic debridement will be performed to treat diseased sites.
  Interventions: Dietary Supplement: Omega-3 polyunsaturated fatty acids; Drug: Aspirin; Procedure: Full-mouth ultrasonic debridement

INTERVENTIONS:
Dietary Supplement: Omega-3 polyunsaturated fatty acids — 3 g of omega-3 polyunsaturated fatty acids daily supplementation over a period of 180 days
  Other Names: Fish oil
  Arms: Test Group
Drug: Aspirin — 100 mg of aspirin daily supplementation over a period of 180 days
  Other Names: acetylsalicylic acid
  Arms: Test Group
Other: Placebo — Placebo pills over a period of 180 days
  Arms: Control group
Procedure: Full-mouth ultrasonic debridement — Full-mouth ultrasonic debridement will be performed in order to treat diseased sites
  Other Names: Periodontal debridement

SUMMARY:
The aim of this randomized controlled clinical trial of superiority will be to evaluate the effect of 3 g of omega-3 polyunsaturated fatty acids and 100 mg of aspirin daily supplementation over a period of 180 days as adjunct to non-surgical therapY of patients with generalized aggressive periodontitis. Probing depth, clinical attachment level, gingival index and concentration of microorganisms and cytokines at baseline, 3, and 6 12 months after the procedure will be evaluated.

DETAILED DESCRIPTION:
The study methodology is according to CONSORT-STATEMENT 2010 for randomized controlled clinical trials.

Study Design The study is designed as a prospective, interventional, parallel, blinded, randomized, controlled clinical trial of superiority.

Source of data The population of this study will be recruited among patients referred to the Science and Technology Institute - ICT- São José dos Campos, College of Dentistry. Patients will fill a healthy history questionnaire to ensure that they are medically qualified for participate in this study. Based on the power calculation for this study, a population of 38 patients will be included. Considering α of 5% and 10% β-type error (90% power) to detect a difference of at least 1 mm in probing depth reduction of pockets ≥ 5 mm between groups, for a standard deviation of 0.94 from a previous study evaluating different antimicrobials in the treatment of GAgP (Xajigeorgiou et al., 2006), 19 patients will be needed in each group.

Clinical Parameters All clinical parameters will be assessed by a single blinded, trained and calibrated examiner (CFA) before periodontal therapy (baseline) and at 3 and 6 months after using a manual probe. Measurements will be done at six sites per tooth (mesiobuccal, buccal, disto-buccal, distolingual, lingual, and mesiolingual) in all teeth, except third molars.

The following clinical parameters will be evaluated: 1) Full-mouth plaque index (FMPI); 2) Bleeding on probing (BoP); 3) Probing depth (PD): distance from the bottom of sulcus/pocket to gingival margin; 4) Gingival recession (GM): distance from the free gingival margin to cement-enamel junction (CEJ); 5) Clinical attachment level (CAL): distance from bottom of sulcus/pocket to the CEJ. The CEJ will be identified by careful probe on cervical area.

Calibration and Randomization Initially, a total of ten patients presenting with GAgP will be selected. The designated examiner (CFA) will measure CAL and PD in all patients twice within 24 hours, with an interval of ≥ 1 hour between examinations. Then, the measures will be submitted to intraclass correlation test and the examiner will be judged calibrated if reaches 90% agreement.

Patients will be allocated into two groups according to a computer-generated list. The allocation will be implemented by an investigator (NC) who was not directly involved in the examination or treatment procedures.

Treatment Protocols

All patients will be treated with periodontal therapy through of the one-stage, full mouth, ultrasonic debridement (FMUD). In a single session, patients will receive local anesthesia and periodontal debridement with ultrasound equipment (Cavitron - Dentsply EUA) and subgingival tips (UI25KSF10S, Hu-Friedy). All diseased sites will be instrumented in this one session. The debridement session will be performed by a single experienced and trained periodontist (NA), different from the examiner. Immediately before the mechanical therapy, patients will be allocated in one of the two treatment protocols:

Test group (n = 19): FMUD + 3 g of omega-3 polyunsaturated fatty acids and 100 mg of aspirin daily supplementation over a period of 180 days; Control group (n = 19): FMUD + placebo pills.

All patients will start taking the pills immediately before of the FMUD session.

Microbiological evaluation Subgingival microbiological samples will be collected at the baseline, 3 and 6 months after therapy. The site will be isolated with a sterile cotton roller and supragingival biofilm will be carefully removed with periodontal curettes and a sterile paper will be inserted into the periodontal pocket for 30 s (Hartoth et al., 1999). The sample will be stored in sterile microtubes. The samples will then be lyophilized and sent to the Department of Periodontology at the University of Florida, where the samples will be analyzed.

Evaluation of cytokines For the analysis of immunological changes, crevicular gingival fluid (CGF) will be collected at baseline, 3 and 6 months after treatment. Each site will be isolated with a sterile cotton roller and the supragingival biofilm will be removed. After this, the CGF will be collected with Periopaper strips (Periopaper, Oraflow, Plainview, NY, USA), inserted in the pocket for 15 seconds. The volume of collected fluid will be measured (Periotron 8000, Oraflow). The Periopaper strips will be stored in a sterile tube containing 300μl of phosphate saline (PBS) with 5% Tween-20 and stored in a freezer at -20 ° C until the multiplex test. The level of the following cytokines will be measured in the CGF: interferon (IFN) -γ, interleukins (IL) -10, -1β, -4, -6, -8, tumor necrosis factor (TNF) -α, macrophage inflammatory protein 1α (MIP1α), 1α monocyte chemotactic protein (MCP-1α). The 10-plex high sensitivity kit (Millipore Corporation, Billerica, MA, USA) will be used according to the manufacturer's instruction and analyzed using the MAGpixTM platform (MiraiBio, Alameda, CA, USA). Samples will be analyzed individually (each pocket separately) and the concentrations will be calculated using a standard 5-parameter curve in the Xponet program (Millipore Corporation). The concentration of each marker will be given in pg / ml. All analysis of cytokine concentrations will be done in duplicate.

Statistical analysis Two analyzes will be performed: Per Protocol and Intention-to-treat (Moher, 2010; Gupta, 2011; Day, 2008). For each of them, mean and standard deviation will be calculated in each of the parameters. Full-mouth PI, GI, PD, CAL, and GR will be submitted to the Shapiro-Wilk test to evaluate the distribution of these data, and then subjected to the variance test for both intra- and intra-group comparison. In addition, the number of pockets ≥ 5mm, the frequency of closure of these pockets, the mean reduction in PS and the gain in CAL of these pockets will be assessed before and after the therapy by performing intra- and inter-group analyzes.

The concentration of each cytokine will be analyzed by test of variance for intra and intergroup comparison.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of GAgP (AAP, 1999);
* presence of ≥20 teeth;
* presence of ≥ 6 sites presenting PD ≥ 5mm with bleeding on probing (BOP) and ≥2 sites with PD ≥7mm (including incisors and first molars, in addition to other two non-contiguous teeth);
* good general health;
* agree to participate in the study and sign a written informed consent. All subjects will be individually informed about the objectives, probable risks and benefits of the protocol treatment (according to Resolution nº196 of October 1996 and to the Professional Code of Dental Ethics - 179/93).

Exclusion Criteria:

* pregnancy or lactating;
* suffer from any systemic disease (e.g. cardiovascular disorders, diabetes, blood dyscrasias, immunodeficiency, etc) which could alter the course of periodontal disease;
* took antimicrobials in the previous 6 months;
* taking long-term anti-inflammatory drugs;
* previous periodontal treatment within the last 12 months;
* smoker ≥ 10 cigarettes.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Santamaria, Professor, Principal Investigator — Universidade Estadual Paulista "Julio de Mesquita Filho", ICT/UNESP
Locations (1):
- College of Dentistry - São José dos Campos, Sao Paulo State University, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-Sharkawy H, Aboelsaad N, Eliwa M, Darweesh M, Alshahat M, Kantarci A, Hasturk H, Van Dyke TE. Adjunctive treatment of chronic periodontitis with daily dietary supplementation with omega-3 Fatty acids and low-dose aspirin. J Periodontol. 2010 Nov;81(11):1635-43. doi: 10.1902/jop.2010.090628. Epub 2010 Jun 23. PMID 20572767

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: In this group (n = 19), patients took placebo pills and full-mouth ultrasonic debridement was performed to treat diseased sites.
  Placebo: Placebo pills over a period of 180 days
  Full-mouth ultrasonic debridement: Full-mouth ultrasonic debridement will be performed in order to treat diseased sites
- Test Group: In this group (n = 19), patients took 900 mg of omega-3 polyunsaturated fatty acids and 100 mg of aspirin daily over a period of 180 days and full-mouth ultrasonic debridement was performed to treat diseased sites.
  Omega-3 polyunsaturated fatty acids: 900 mg of omega-3 polyunsaturated fatty acids daily supplementation over a period of 180 days
  Aspirin: 100 mg of aspirin daily supplementation over a period of 180 days
  Full-mouth ultrasonic debridement: Full-mouth ultrasonic debridement will be performed in order to treat diseased sites
Period: Overall Study
Arm/Group | Control Group | Test Group
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Group: In this group (n = 19), patients received placebo pills over a period of 180 days and full-mouth ultrasonic debridement was performed to treat diseased sites.
- Test Group: In this group (n = 19), patients received 900 mg of omega-3 polyunsaturated fatty acids and 100 mg of aspirin daily over a period of 180 days and full-mouth ultrasonic debridement was performed to treat diseased sites.
- Total: Total of all reporting groups
Arm/Group | Control Group | Test Group | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.42 (5.79) | 32.84 (5.47) | 31.63 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 5 | 7 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change in Probing Depth
Description: Evaluate the difference between baseline and 6 months PD measures.
Time Frame: Baseline, 3 and 6 months
Measure: Mean (Standard Deviation); unit: milimeters
Groups:
- Control Group: In this group (n = 19), patients took placebo pills over a period of 180 days and received full-mouth ultrasonic debridement to treat diseased sites.
- Test Group: In this group (n = 19), patients will take 900 mg of omega-3 polyunsaturated fatty acids and 100 mg of aspirin daily over a period of 180 days and full-mouth ultrasonic debridement was performed to treat diseased sites.
Arm/Group | Control Group | Test Group
Number analyzed (Participants) | 19 | 19
milimeters
  Baseline | 3.88 (0.15) | 3.74 (0.15)
  3 months | 3.38 (0.14) | 3.26 (0.13)
  6 months | 3.37 (0.14) | 3.25 (0.13)
Statistical Analysis 1: Comparison: Control Group vs Test Group; Test type: Superiority; p < 0.05, Generalized Estimated Equations

2. Secondary Outcome: Change in Clinical Attachment Level
Description: Evaluate the difference between baseline and 6 months CAL measures.
Time Frame: Baseline, 3 and 6 months
Measure: Mean (Standard Deviation); unit: milimeters
Arm/Group | Control Group | Test Group
Number analyzed (Participants) | 19 | 19
milimeters
  Baseline | 3.94 (0.17) | 4.01 (0.21)
  3 months | 3.58 (0.17) | 3.65 (0.21)
  6 months | 3.59 (0.17) | 3.64 (0.2)
Statistical Analysis 1: Comparison: Control Group vs Test Group; Test type: Superiority; p < 0.05, Generalized Estimated Equations

3. Secondary Outcome: Change in Bleeding on Probe
Description: Evaluate the difference between baseline and 6 months BoP measures
Time Frame: Baseline, 3 and 6 months
Measure: Mean (Standard Deviation); unit: percentage of sites with BoP
Arm/Group | Control Group | Test Group
Number analyzed (Participants) | 19 | 19
percentage of sites with BoP
  Baseline | 54.11 (4.97) | 44.58 (3.72)
  3 months | 33.27 (3.72) | 27.41 (2.35)
  6 months | 31.77 (3.58) | 26.17 (2.18)
Statistical Analysis 1: Comparison: Control Group vs Test Group; Test type: Superiority; p < 0.05, Generalized Estimated Equations

ADVERSE EVENTS:
Time Frame: During 6 months
Arm/Group | Control Group | Test Group
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-22): https://cdn.clinicaltrials.gov/large-docs/46/NCT03093246/Prot_SAP_000.pdf